CLINICAL TRIAL: NCT01939821
Title: A Pilot Study to Evaluate Feasibility of Educational Programs With Regard to Good Fecal Incontinence Care in Nursing Homes
Brief Title: A Pilot Study to Evaluate Educational Programs to Improve Fecal Incontinence Care in Nursing Homes
Acronym: PEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HIST; ES507368 (Other: Sør-Trøndelag University College, Norway)
Record Dates: First submitted 2013-07-04; First posted 2013-09-11 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Fecal Incontinence; Staffs' Attitudes
Keywords: Fecal incontinence; attitudes; knowledge; quality of care
MeSH Terms: conditions — Fecal Incontinence; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Educational and counselling program (Experimental): In addition to educational meeting and printed educational material the investigators will include the use of local opinion leaders and educational outreach
  Interventions: Behavioral: Educational and counselling program
- Educational program (Active Comparator): The investigators want to organize the educational meetings as an interactive workshop that target knowledge, attitudes, and skills at the individual healthcare professional/peer group level.
  Interventions: Behavioral: Educational program
- Control group (No Intervention): The control group will not receive any educational program. It represents the present real life in nursing homes.

INTERVENTIONS:
Behavioral: Educational and counselling program — Educational and counselling program: In addition to educational meeting and printed educational material the investigators will include the use of local opinion leaders and educational outreach . Local opinion leaders are defined as "use of providers nominated by their colleges as educationally influential". Opinion leadership is the degree to which an individual is able to influence other individual's attitudes or overt behavior informally in a desired way with relative frequency. Educational outreach is defined as "use of a trained person who meets with providers in their practice setting to give information with the intent of changing the providers practice."
  Arms: Educational and counselling program
Behavioral: Educational program — Educational program: Educational meeting and printed educational material Educational meeting is defined as "participation of healthcare providers in conference, lectures, workshops or traineeships". The investigators want to organize the educational meetings as an interactive workshop that target knowledge, attitudes, and skills at the individual healthcare professional/peer group level. Printed educational material is defined as "distribution of published or printed recommendations for clinical care, including clinical practice guidelines". In general, printed educational material target knowledge and potential skill gaps of individual healthcare professionals.
  Arms: Educational program

SUMMARY:
The investigators are planning to do a cluster randomized trial to test the effect of different educational programs for staff according to nursing home patients FI (fecal incontinence). Since there are very few published trials of treatment of FI in older people, and no rigorously evaluated studies on interventions for FI in nursing homes, or rigorously evaluated continence education program for staff concerning continence care, a pilot study is necessary. The aim for the pilot study is to evaluate feasibility, acceptability and adherence according to the educational intervention, methods used and outcome measures. This is designed to be an external pilot study. External pilot studies are small scale versions of the main study which are not intended to be part of the main study. The pilot intervention period is 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes Wards with 24 hour long term care residency, similar nurse/patient ratio and General Practitioner consultancy, comparable patient groups according to frailty, comparable ward size according to number of patients and staff.
* Patients All patients on long term residency (1 month or more) are eligible for measurements.
* Registered nurses (RN) and authorized social educators (ASE) RN's and ASE's with position above 50% are eligible according to participation in the educational meeting and to be recruited as a local opinion leader in intervention 2. All staff is invited to the educational outreach meetings throughout the intervention period.

Exclusion Criteria:

* Nursing homes with diverse staff and patient composition
* Patients on short term residency
* Registered nurses (RN) and authorized social educators (ASE) RN's and ASE's with position less than 50%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The proportion patients assessed by the clinical guidelines | 3 months
  90% of the patients assessed by the clinical guideline

SECONDARY OUTCOMES:
Proportion of completed patient health questionnaires | 3 months
  Response rate more than 80%
Acceptable performance of multiple choice test measuring change in staff knowledge. | 3 months
  80% claim that the test set understandable and relevant
The proportion of missing data in each completed questionnaire | 3 months
  Less than 10%

CONTACTS AND LOCATIONS:
Overall Officials: Lene Blekken, DrPH, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Sør-Trøndelag University College, Trondheim, Norway

REFERENCES:
- [Result] Blekken LE, Nakrem S, Gjeilo KH, Norton C, Morkved S, Vinsnes AG. Feasibility, acceptability, and adherence of two educational programs for care staff concerning nursing home patients' fecal incontinence: a pilot study preceding a cluster-randomized controlled trial. Implement Sci. 2015 May 23;10:72. doi: 10.1186/s13012-015-0263-8. PMID 26002520